CLINICAL TRIAL: NCT00128427
Title: Treatment and Prevention of Pericarditis With Colchicine. A Multicenter Double Blind Randomized Trial. The COPPS Trial: COlchicine for the Prevention of Postpericardiotomy Syndrome
Brief Title: Study of Colchicine to Prevent the Postpericardiotomy Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Sanitaria Locale 3, Torino (Other)
Responsible Party: Azienda Sanitaria Locale 3, Torino, Ospedale Maria Vittoria, Torino
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DCASL30501-3; EUDRACT number 2005-001570-28
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Postpericardiotomy Syndrome
Keywords: Postpericardiotomy Syndrome; Pericarditis; Prevention; Colchicine; Recurrence
MeSH Terms: conditions — Postpericardiotomy Syndrome; Pericarditis; Recurrence | interventions — Colchicine; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Colchicine (for 1 month)

SUMMARY:
The purpose of the study is to determine whether colchicine is safe and effective in the prevention of the postpericardiotomy syndrome.

DETAILED DESCRIPTION:
The postpericardiotomy syndrome is a frequent complication after cardiac surgery affecting from 20 to 40% of patients. The etiology of this complication is a subject of debate. It is commonly believed to be an autoimmune response to pericardial and/or pleural bleeding or surgical trauma. Colchicine is safe and effective in the treatment and prevention of pericarditis and preliminary data have shown that it may be effective also in the primary prevention of the postpericardiotomy syndrome.

Comparisons: The study will compare the safety and efficacy of colchicine in the primary prevention of the postpericardiotomy syndrome in addition to optimal standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the third day after a cardiac surgery operation
* Age≥ 18 years
* Informed consent

Exclusion Criteria:

All evaluated before the surgical operation:

* Known severe liver disease and/or elevated transaminases >1.5 times the upper limit of normality
* Serum creatinine >2.5 mg/dl
* Serum creatine kinase (CK) over the upper limit of normality or known myopathy
* Known gastrointestinal or blood disease
* Pregnant or lactating women or women not protected by a contraception method
* Known hypersensibility to colchicine
* Treatment with colchicine at enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Postpericardiotomy syndrome | 12 months

SECONDARY OUTCOMES:
Disease-related hospitalization, cardiac tamponade, constrictive pericarditis and relapses

CONTACTS AND LOCATIONS:
Overall Officials: Rita TRINCHERO, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital. ASL 3. Torino.; Massimo IMAZIO, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital. ASL 3. Torino.; Massimo IMAZIO, MD, Principal Investigator — Cardiology Department. Maria Vittoria Hospital. ASL 3. Torino.
Locations (6):
- Italy (6):
  - Ospedali Riuniti, Bergamo, Bergamo
  - Ospedale Regionale Bolzano, Bolzano, Bolzano
  - Ospedale Niguarda, Milan, Milano
  - Cardiology Department. Maria Vittoria Hospital. ASL 3. Torino., Torino, Torino
  - Cardiac Surgery- Ospedale Mauriziano, Torino, Torino
  - Ospedale di Rivoli, Rivoli

REFERENCES:
- [Derived] Imazio M, Brucato A, Ferrazzi P, Rovere ME, Gandino A, Cemin R, Ferrua S, Belli R, Maestroni S, Simon C, Zingarelli E, Barosi A, Sansone F, Patrini D, Vitali E, Trinchero R, Spodick DH, Adler Y; COPPS Investigators. Colchicine reduces postoperative atrial fibrillation: results of the Colchicine for the Prevention of the Postpericardiotomy Syndrome (COPPS) atrial fibrillation substudy. Circulation. 2011 Nov 22;124(21):2290-5. doi: 10.1161/CIRCULATIONAHA.111.026153. Epub 2011 Nov 16. PMID 22090167
- [Derived] Imazio M, Brucato A, Rovere ME, Gandino A, Cemin R, Ferrua S, Maestroni S, Zingarelli E, Barosi A, Simon C, Sansone F, Patrini D, Vitali E, Belli R, Ferrazzi P, Trinchero R, Spodick DH, Adler Y. Colchicine prevents early postoperative pericardial and pleural effusions. Am Heart J. 2011 Sep;162(3):527-32.e1. doi: 10.1016/j.ahj.2011.05.017. Epub 2011 Jul 18. PMID 21884871
- [Derived] Imazio M, Trinchero R, Brucato A, Rovere ME, Gandino A, Cemin R, Ferrua S, Maestroni S, Zingarelli E, Barosi A, Simon C, Sansone F, Patrini D, Vitali E, Ferrazzi P, Spodick DH, Adler Y; COPPS Investigators. COlchicine for the Prevention of the Post-pericardiotomy Syndrome (COPPS): a multicentre, randomized, double-blind, placebo-controlled trial. Eur Heart J. 2010 Nov;31(22):2749-54. doi: 10.1093/eurheartj/ehq319. Epub 2010 Aug 30. PMID 20805112